CLINICAL TRIAL: NCT05028335
Title: Effect of 1.5% Potassium Oxalate on the Control of Tooth Sensitivity and Color Change After Home Bleaching: a Randomized, Placebo-controlled Clinical Study
Brief Title: Effect of 1.5% Potassium Oxalate on the Control of Tooth Sensitivity and Color Change After Home Bleaching
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Para (Other)
Responsible Party: Principal Investigator, Cecy Martins Silva, clinical professor, Universidade Federal do Para
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: UFPara-0010
Record Dates: First submitted 2021-08-24; First posted 2021-08-31 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Carbamide Peroxide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group G1 (Other): Home bleaching treatment (Carbamide Peroxide (PC) 22%) + placebo gel
  Interventions: Other: Carbamide Peroxide (PC) 22%) + placebo gel
- Group G2 (Experimental): Home bleaching treatment (Carbamide Peroxide (PC) 22%) + 1.5% Potassium Oxalate gel
  Interventions: Other: Carbamide Peroxide (PC) 22%) + Potassium Oxalate gel 1.5%

INTERVENTIONS:
Other: Carbamide Peroxide (PC) 22%) + placebo gel — Application of one drop of Polanight bleaching agent (SDI, SP, Brazil) on each corresponding tooth in a tray that was used for 45 minutes a day, for a period of twenty-one days. After the bleaching treatment, the participants were instructed to wash the trays under running water and dry them. The volunteers were instructed to apply a small amount of placebo gel, without active ingredient, with color, texture and odor similar to 1.5% oxalate gel (Painless, BM4, SC, Brazil) in the spaces related to the vestibular portions of the teeth trays, which were used for 10 minutes.
  Arms: Group G1
Other: Carbamide Peroxide (PC) 22%) + Potassium Oxalate gel 1.5% — Application of one drop of Polanight bleaching agent (SDI, SP, Brazil) on each corresponding tooth in a tray that was used for 45 minutes a day, for a period of twenty-one days. After the bleaching treatment, the participants were instructed to wash the trays under running water and dry them with absorbent paper. The volunteers applied a small amount of 1.5% potassium oxalate gel (Painless, BM4, SC, Brazil) in the spaces relative to the vestibular portions of the tray's teeth, which were used for 10 minutes.
  Arms: Group G2

SUMMARY:
This double-blind randomized clinical trial evaluated the effect of 1.5% potassium oxalate on pain sensitivity control and color change after home tooth whitening. It also evaluated the influence of potassium oxalate on health-related quality of life (HRQOL) and on the degree of patient satisfaction after bleaching treatment.

ELIGIBILITY:
Inclusion Criteria:

* individuals aged 18 to 29 years of both sexes with chroma greater than A2 in the upper incisors and canines, in the Vita Classical color scale;
* absence of active caries lesions
* patients who had never undergone bleaching therapy;
* good oral hygiene and no hypersensitivity to tactile and evaporative stimuli through the Visual Analog Pain Scale;

Exclusion Criteria:

* patients undergoing fixed orthodontic treatment;
* patients with darkened non-vital teeth and/or with extensive restorations in molars;
* presence of cracks or fractures;
* patients allergic to the product, with the presence of gastroesophageal disorders and with dentinal exposure in anterior and/or posterior teeth.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-06-05 (Actual)

PRIMARY OUTCOMES:
dentin sensitivity | 21 days after the start of the whitening treatment
  evaluation of dentinal sensitivity during treatment through a daily questionnaire, using a visual analogue scale with values from 0 to 10, with higher values indicating a worse level of pain.
dental color assessment | 21 days and 1 month after the bleaching treatment
  Color evaluation was performed using the EasyshadeAdvanced spectrophotometer (Vita-Zahnfabrik, GE, Germany), using the CIE L*a*b* system.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Pará, Belém, Pará, Brazil